CLINICAL TRIAL: NCT07263269
Title: Assessment of Dumping and Quality of Life 6 Months Following Sleeve Gastrectomy With and Without Transit Bipartition : Comparative Study
Brief Title: Comparing Dumping Symptoms and Quality of Life 6 Months After Sleeve Gastrectomy With or Without Transit Bipartition in Adults With Obesity
Acronym: STuD-QoL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mina Kamal Gergis Erian (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Sponsor-Investigator, Mina Kamal Gergis Erian, General and laparoscopic Surgery Specialist, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-109-2024
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Morbid Obesity; Dumping Syndrome; Postgastrectomy Syndrome; Quality of Life; Bariatric Surgery; Metabolic Diseases; Gastrointestinal Function Disorders; Sleeve Gastrectomy; Gastrointestinal Transit; Nutritional Status; Patient-reported Outcome Measures
Keywords: Sleeve Gastrectomy; Transit Bipartition; Bariatric Surgery; Metabolic Surgery; Dumping Syndrome; Postgastrectomy Syndrome; Quality of Life; Obesity; Morbid Obesity; Gastrointestinal Function; Postoperative Complications; Weight Loss Outcomes; Gastrointestinal Transit; Metabolic Outcomes; Patient-Reported Outcomes; Comparative Study
MeSH Terms: conditions — Obesity; Obesity, Morbid; Dumping Syndrome; Postgastrectomy Syndromes; Metabolic Diseases; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve Gastrectomy (LSG) Group (Active Comparator): This group will undergo the standard sleeve gastrectomy (LSG) procedure, where a large portion of the stomach is removed, leaving a tube-like structure. The effects of this procedure on dumping syndrome and quality of life will be assessed and compared to the SG-TB group.
  Intervention: Sleeve gastrectomy surgery (no transit bipartition).
  Interventions: Procedure: Sleeve Gastrectomy
- Sleeve Gastrectomy with Transit Bipartition (SG-TB) Group (Experimental): Participants will undergo sleeve gastrectomy combined with transit bipartition, a modified procedure involving the rerouting of part of the small intestine. Outcomes regarding dumping syndrome and quality of life will be evaluated and compared with the LSG group.
  Interventions: Procedure: Sleeve Gastrectomy with Transit Bipartition

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — Sleeve gastrectomy is a weight loss surgery where approximately 75-80% of the stomach is surgically removed, leaving a narrow, tube-like structure. This reduces the stomach's volume, limiting food intake, and promoting weight loss. It is often performed laparoscopically and requires no rerouting of the intestines. The procedure is commonly used to treat morbid obesity and related metabolic conditions.
  Arms: Sleeve Gastrectomy (LSG) Group
Procedure: Sleeve Gastrectomy with Transit Bipartition — This modified version of sleeve gastrectomy involves both the removal of a large portion of the stomach and the rerouting of a part of the small intestine (transit bipartition). This alteration changes the gut hormone response, potentially reducing the risk of dumping syndrome and improving metabolic outcomes. Like LSG, it is typically performed laparoscopically and focuses on both weight loss and gastrointestinal function modification.
  Arms: Sleeve Gastrectomy with Transit Bipartition (SG-TB) Group

SUMMARY:
This clinical study aims to compare two types of bariatric (weight loss) surgery used to treat obesity: sleeve gastrectomy alone and sleeve gastrectomy with transit bipartition. Both procedures help patients lose excess weight and improve obesity-related conditions such as diabetes and high blood pressure. However, they may differ in how they affect digestion and patients' quality of life after surgery.

One possible complication after bariatric surgery is dumping syndrome. This occurs when food passes too quickly from the stomach into the small intestine, causing symptoms such as nausea, bloating, abdominal pain, diarrhea, dizziness, or fatigue after eating. These symptoms can be uncomfortable and may interfere with daily activities, eating habits, and overall well-being.

The main goal of this study is to evaluate and compare both the occurrence of dumping syndrome and the overall quality of life six months after surgery in two groups of patients:

Those who undergo sleeve gastrectomy alone.

Those who undergo sleeve gastrectomy combined with transit bipartition.

Participants will be adults with obesity who are scheduled to undergo bariatric surgery. Each participant will be evaluated before and after surgery using medical assessments and validated questionnaires that measure symptoms, eating patterns, and different aspects of quality of life-including physical health, emotional well-being, and social functioning.

Follow-up visits and questionnaires will be conducted six months after surgery to determine how each surgical technique affects patients' digestion, comfort after meals, and overall satisfaction with their health and lifestyle.

The study's hypothesis is that adding transit bipartition to sleeve gastrectomy may decrease the frequency or severity of dumping syndrome and lead to better quality of life outcomes compared to sleeve gastrectomy alone.

By comparing these two surgical approaches, this study hopes to help surgeons and patients make better-informed decisions about bariatric surgery, aiming for the best combination of effective weight loss, minimal side effects, and improved long-term quality of life.

DETAILED DESCRIPTION:
Background and Rationale

Obesity has become one of the most important public-health challenges worldwide. It is associated with a wide range of comorbid conditions such as type 2 diabetes mellitus, hypertension, dyslipidemia, non-alcoholic fatty liver disease, obstructive sleep apnea, degenerative joint disease, and increased cardiovascular morbidity and mortality. Conservative management strategies-including dietary modification, physical activity, and pharmacologic therapy-often result in only modest and temporary weight reduction. Consequently, bariatric and metabolic surgery has emerged as the most effective and durable intervention for achieving long-term weight loss and improvement or remission of obesity-related diseases.

Among the different bariatric procedures, laparoscopic sleeve gastrectomy (LSG) has gained worldwide popularity. It is technically simpler than gastric bypass procedures and does not involve intestinal anastomoses or foreign materials. During LSG, approximately 75-80% of the stomach is resected along the greater curvature, leaving a tubular gastric "sleeve." This results in restrictive limitation of food intake and favorable hormonal changes, such as decreased ghrelin secretion, leading to appetite suppression. LSG has proven effective in producing substantial and durable weight loss as well as improvement in metabolic parameters.

However, despite these benefits, some patients experience functional gastrointestinal symptoms after LSG, including gastroesophageal reflux disease, food intolerance, early satiety, and dumping syndrome. Dumping syndrome refers to a collection of symptoms that occur when food passes too rapidly from the stomach into the small intestine. It can be divided into early dumping (occurring 10-30 minutes after eating, with symptoms such as nausea, abdominal cramps, palpitations, and dizziness) and late dumping (1-3 hours after eating, characterized by hypoglycemia, fatigue, and sweating). These symptoms may significantly impair quality of life (QoL), limit dietary freedom, and affect social activities.

To enhance the metabolic efficacy of sleeve gastrectomy while minimizing complications, several hybrid or modified techniques have been introduced. One such modification is sleeve gastrectomy with transit bipartition (SG-TB). In this operation, a side-to-side anastomosis is created between the distal ileum and the antrum or the first portion of the duodenum, allowing ingested food to pass through both the natural duodenal route and an alternative shortcut to the distal small intestine. This design maintains continuity of the biliary and pancreatic secretions, preserves access to the duodenum for endoscopy, and reduces the risk of nutritional deficiencies commonly seen with complete bypass procedures. Physiologically, the presence of dual intestinal transit is believed to enhance incretin hormone release (GLP-1, PYY) and improve insulin sensitivity.

Although previous studies have demonstrated that SG-TB can achieve excellent weight loss and glycemic control, comparative data regarding postoperative functional symptoms and QoL outcomes remain limited. Because dumping syndrome and related symptoms can significantly affect patient satisfaction and long-term adherence to dietary recommendations, it is essential to understand whether the addition of transit bipartition alters these outcomes relative to the standard sleeve gastrectomy.

Objectives

Primary Objective:

To compare the incidence and severity of dumping syndrome at six months after surgery between patients undergoing sleeve gastrectomy (LSG) and those undergoing sleeve gastrectomy with transit bipartition (SG-TB).

Secondary Objectives:

To compare quality of life (QoL) scores between both groups using validated QoL questionnaires specific to bariatric and gastrointestinal surgery.

To evaluate weight loss outcomes (percentage of excess weight loss, change in body mass index).

To assess improvement or remission of metabolic comorbidities (type 2 diabetes, hypertension, dyslipidemia).

To analyze nutritional and biochemical parameters (iron, vitamin B12, folate, calcium, albumin).

To record and compare postoperative complications and re-intervention rates.

Hypothesis

The study hypothesizes that adding transit bipartition to sleeve gastrectomy will reduce the frequency and/or severity of dumping syndrome by preserving a more physiologic gastric emptying mechanism and offering dual pathways for food transit. Additionally, the hormonal and metabolic benefits of SG-TB are expected to result in improved overall quality of life compared with standard sleeve gastrectomy at six months postoperatively.

Study Design

This is a prospective, comparative, single-center (or multicenter, if applicable) clinical study involving two parallel groups of adult patients undergoing bariatric surgery for the management of obesity.

Group A: Laparoscopic sleeve gastrectomy (LSG)

Group B: Laparoscopic sleeve gastrectomy with transit bipartition (SG-TB)

Patients will be evaluated preoperatively and followed for at least six months after surgery. Allocation to surgical technique will depend on preoperative multidisciplinary assessment and patient-surgeon agreement. All procedures will be performed by experienced bariatric surgeons following standardized techniques to minimize operative variability.

Study Population

Eligible participants will include adult men and women aged 18-60 years with a body mass index (BMI) ≥ 35 kg/m² with comorbidities, or ≥ 40 kg/m² regardless of comorbidities, who are candidates for bariatric surgery according to international guidelines. All participants must be willing to comply with postoperative follow-up visits and to complete the required questionnaires. Exclusion criteria (listed elsewhere in the protocol) include previous major gastric surgery, significant psychiatric illness, pregnancy, or inability to provide informed consent.

Preoperative Evaluation

Before surgery, all participants will undergo:

Full medical history and physical examination

Anthropometric measurements (weight, height, BMI, waist circumference)

Laboratory investigations (complete blood count, liver and renal function, fasting glucose, lipid profile, HbA1c, vitamins and micronutrients)

Assessment of comorbidities

Baseline quality of life assessment using standardized questionnaires (e.g., Gastrointestinal Quality of Life Index (GIQLI), Bariatric Analysis and Reporting Outcome System (BAROS), or SF-36)

Documentation of eating habits and gastrointestinal symptoms

Surgical Technique Overview

Laparoscopic Sleeve Gastrectomy (LSG):

Performed using 4-5 ports under general anesthesia. The greater curvature of the stomach is mobilized starting approximately 4-6 cm from the pylorus up to the angle of His. A 36-40 French calibration tube is used to guide gastric transection with linear staplers, creating a narrow gastric sleeve. The resected stomach is removed, and staple lines are inspected for bleeding or leakage.

Sleeve Gastrectomy with Transit Bipartition (SG-TB):

The sleeve component is created as described above. In addition, a side-to-side anastomosis is fashioned between the distal ileum (typically 250 cm from the ileocecal valve) and the antrum or first part of the duodenum, allowing a dual pathway of food transit. The mesenteric defect is closed to prevent internal herniation. This configuration aims to enhance incretin secretion and glycemic control without complete exclusion of the duodenum.

All operations will be performed laparoscopically. Standardized postoperative protocols for pain management, diet progression, and nutritional supplementation will be applied to both groups.

Postoperative Follow-Up and Assessments

Patients will be followed at regular intervals-typically at 1 month, 3 months, and 6 months postoperatively-with longer follow-up continuing as per institutional policy.

Clinical and Functional Evaluation:

Measurement of weight, BMI, and percentage of excess weight loss (%EWL)

Monitoring of vital signs and comorbid disease status

Documentation of postoperative complications (leak, bleeding, infection, bowel obstruction)

Dumping Syndrome Assessment:

At each follow-up visit, patients will be screened for dumping symptoms using a standardized questionnaire and scoring system, such as the Sigstad Diagnostic Index or Arts Dumping Score. The frequency, severity, and timing of symptoms (early vs. late dumping) will be recorded.

Quality of Life Assessment:

QoL will be evaluated preoperatively and six months postoperatively using validated instruments. Tools may include:

GIQLI (Gastrointestinal Quality of Life Index) - assessing physical, emotional, and social aspects of gastrointestinal health.

BAROS (Bariatric Analysis and Reporting Outcome System) - integrating weight loss, comorbidity resolution, and quality of life changes.

SF-36 Health Survey - measuring overall physical and mental health domains. Patients will complete these questionnaires independently, assisted by study staff if necessary.

Laboratory and Nutritional Monitoring:

Periodic laboratory tests will evaluate glycemic control (fasting glucose, HbA1c), lipid profile, liver function, and micronutrient status (iron, calcium, vitamin B12, folate, vitamin D). Nutritional counseling and supplementation will be provided as per standard bariatric guidelines.

Data Collection and Statistical Analysis

Data will be collected prospectively and entered into a secure database. Continuous variables (e.g., BMI, QoL scores) will be presented as mean ± standard deviation and compared between groups using independent-samples t-tests or Mann-Whitney U tests as appropriate. Categorical variables (e.g., presence of dumping syndrome) will be compared using chi-square or Fisher's exact tests. Within-group comparisons (pre- vs. postoperative) will use paired tests. A p-value < 0.05 will be considered statistically significant.

Multivariate analysis may be used to control for potential confounders such as age, gender, baseline BMI, and presence of diabetes. Correlations between weight loss, dumping score, and QoL improvement will also be explored.

Ethical Considerations

The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. Approval will be obtained from the local Institutional Review Board or Ethics Committee before patient enrollment. All participants will provide written informed consent after being fully informed about the purpose, procedures, potential risks, and benefits of the study. Data confidentiality and patient privacy will be maintained throughout.

Expected Outcomes and Significance

This research is expected to provide a clearer understanding of the functional and quality-of-life outcomes after two common bariatric surgical strategies. Specifically, the study aims to determine whether the addition of transit bipartition to sleeve gastrectomy reduces the incidence of dumping syndrome without compromising weight loss or safety.

If the hypothesis is confirmed, SG-TB may offer a valuable alternative for patients seeking effective metabolic results with fewer functional limitations and better postoperative comfort. Improved quality of life following bariatric surgery is a key determinant of long-term success, patient satisfaction, and adherence to healthy lifestyle changes.

Ultimately, the findings of this comparative study may assist surgeons and multidisciplinary teams in selecting the most appropriate bariatric procedure based on patient characteristics, metabolic goals, and desired postoperative quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI exceeding 40 kg/m2
* BMI exceeding 35 kg/m2, when diagnosed with obesity-related diseases, including type 2 diabetes, hypertension, lipid disorders, and obstructive sleep apnea.
* Obtain informed written consent from the patients or their first guardians
* Patients choosing LSG or LSTB after being offered all suitable bariatric procedures

Exclusion Criteria:

* Patients or their first guardians refusing to participate in the current study.
* Previous bariatric surgeries

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dumping Syndrome | 6 months
  he primary outcome measure is the incidence of dumping syndrome, assessed through patient-reported symptoms and clinical evaluation. Dumping syndrome is characterized by symptoms like nausea, diarrhea, and dizziness that occur after eating, primarily due to rapid gastric emptying.
Quality of Life Assessment | 6 months following surgery
  The quality of life will be assessed using a validated questionnaire, such as the Short Form 36 (SF-36) or Gastrointestinal Quality of Life Index (GIQLI), focusing on physical, emotional, and social well-being. These tools evaluate how the participants feel about their overall health, function, and the impact of their surgery. Key factors include general health perceptions, physical functioning, pain, emotional well-being, and social interactions.

SECONDARY OUTCOMES:
Percentage of Excess Weight Loss (EWL) | 6 months post-surgery
  The percentage of excess weight loss will be measured using the Excess Weight Loss (EWL) formula, which compares the patient's weight loss to their ideal body weight. This metric evaluates the effectiveness of the surgery in achieving weight loss.
Incidence of Surgical Complications | 6 months post-surgery
  This secondary outcome will track any complications arising from the surgery, such as infection, bleeding, leakage, and other post-operative issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berg P, McCallum R. Dumping Syndrome: A Review of the Current Concepts of Pathophysiology, Diagnosis, and Treatment. Dig Dis Sci. 2016 Jan;61(1):11-8. doi: 10.1007/s10620-015-3839-x. Epub 2015 Sep 22. PMID 26396002